CLINICAL TRIAL: NCT00177944
Title: Invasive Fungal Infections Surveillance Initiative
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB # 0503062
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Fungal Infection
Keywords: invasive fungal infection
MeSH Terms: conditions — Mycoses; Invasive Fungal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- patients with funal infections

SUMMARY:
The purpose of this study is to optimize the management of patients treated for invasive fungal infections by establishing a real-time, continuous clinical data base that will capture and monitor trends in the epidemiology, diagnosis, treatment and outcomes of invasive fungal infections; reflect routine clinical management of patients with invasive fungal infections in order to evaluate treatment and provide a rationale for future treatment paradigms; and allow physicians to assess adherence to institutional clinical practice guidelines, validate current standardized definitions for patients with invasive fungal infections and promote change where appropriate.

DETAILED DESCRIPTION:
Gender, height, weight, ethnicity, antifungal treatment, fungal colonization, laboratory results, past medical history, invasive fungal infection diagnosis, medications, outcomes

ELIGIBILITY:
Inclusion Criteria:

* All patients with a diagnosis of proven or probable invasive fungal infection . This includes patients with proven or probable invasive mold infections as well as patients with proven candidemia.

Exclusion Criteria:

* All patients with a diagnosis of possible invasive fungal infection . This includes patients with possible mold infections as well as patients with possible candidemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with funal infections
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2005-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
outcome after invasive fungal infection | 60 days post infection
  outcome after invasive fungal infection

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda Silveira, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States